CLINICAL TRIAL: NCT02683941
Title: A Phase 3, Prospective, Randomized, Double-blind, Multi-center Study of the Efficacy and Safety of Lanreotide Autogel®/Depot 120 mg Plus BSC vs. Placebo Plus BSC for Tumour Control in Subjects With Well Differentiated, Metastatic and/or Unresectable, Typical or Atypical, Lung Neuroendocrine Tumours
Brief Title: Efficacy and Safety of Lanreotide Autogel/ Depot 120 mg vs. Placebo in Subjects With Lung Neuroendocrine Tumours
Acronym: SPINET
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: National Comprehensive Cancer Network & European Neuroendocrine Tumor Society guidelines (2015/2016) led to prescription of somatostatin analogues (SSAs) in this setting, thereby limiting recruitment.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-US-52030-328; 2015-004992-62 (EudraCT Number)
Record Dates: First submitted 2015-09-21; First posted 2016-02-17 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Neuroendocrine Tumors in Lung
MeSH Terms: interventions — lanreotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lanreotide (Autogel formulation) (Experimental): 120mg every 28 days until disease progression, death, or unacceptable toxicity
  Interventions: Drug: Lanreotide (Autogel formulation); Drug: Best Supportive Care
- Placebo (Placebo Comparator): 120mg every 28 days until disease progression, death, or unacceptable toxicity during the double-blind phase. The patient may enter open-label phase for treatment with Lanreotide.
  Interventions: Drug: Placebo; Drug: Best Supportive Care

INTERVENTIONS:
Drug: Lanreotide (Autogel formulation) — 120mg every 28 days until disease progression, death, or unacceptable toxicity
  Other Names: Lanreotide Depot (US)
  Arms: Lanreotide (Autogel formulation)
Drug: Placebo — Saline solution 0.9% administered via deep subcutaneous injection every 28 days until disease progression.
  Arms: Placebo
Drug: Best Supportive Care — Best Supportive Care is best available therapy at the choice of the investigator
  Other Names: BSC

SUMMARY:
This is a Phase 3, prospective, multi-center, randomized, double-blind, study evaluating the efficacy and safety of LAN plus BSC versus placebo plus BSC for the treatment of well-differentiated, metastatic and/or unresectable, typical or atypical bronchopulmonary NETs.

This study contains two phases: the Double-Blind (DB) Phase, and the Open Label (OL) Phase. The DB Phase includes: Screening, Baseline and Treatment period. The OL Phase will consist of two periods: Treatment Period and Follow-Up Period.

The primary objective will be to describe the antitumour efficacy of Lanreotide Autogel/Depot 120 mg (LAN) plus Best Supportive Care (BSC) every 28 days, in terms of progression-free survival (PFS), measured by central review using Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 criteria, every 12 weeks, in subjects randomized to LAN with unresectable and/or metastatic well differentiated, typical or atypical bronchopulmonary neuroendocrine tumours.

Recent updates of National Cancer Institute Cancer Network (NCCN) & European Neuroendocrine Tumor Society (ENETS) guidelines recommend SSA in first line for the treatment of locoregional unresectable or metastatic bronchopulmonary NETs as an option beyond 'observation' leading to slow and difficult recruitment in SPINET study. Consequently, it was decided to prematurely stop the recruitment in the SPINET study and to transition all subjects still treated in the double-blind phase to the open label (OL) treatment and follow-up phases following respective country approvals of Amendment #5.

The new aim of this Phase 3, multicenter, prospective, randomized placebo-controlled clinical study is to describe the antitumor efficacy and safety of Lanreotide Autogel/Depot 120 mg (LAN) plus Best Supportive Care (BSC) in subjects with well-differentiated, metastatic and/or unresectable, typical or atypical, bronchopulmonary NETs.

DETAILED DESCRIPTION:
As planned initially, a total of 216 eligible patients with well-differentiated typical or atypical, metastatic and/or unresectable bronchopulmonary NETs, and a positive somatostatin receptor imaging (SRI) (Octreoscan® ≥ grade 2 Krenning scale; Ga-PET scan: uptake greater than liver background), were to be randomized 2:1 to either LAN plus BSC (120mg/28 days) or placebo plus BSC following the stratification of 1) typical versus atypical and 2) prior chemotherapy versus no prior chemotherapy*.

* cytotoxic chemotherapy or molecular targeted therapy or interferon.

At the time of the premature stop of the recruitment (as per Protocol Amendment #5), 77 patients were enrolled. All patients still treated in the DB Phase were entered into the OL Phase (either for Follow up or for OL treatment periods). The transition to the OL periods was done on a country-basis and per patient, at the following planned scheduled visit (i.e. approximately 28 days from the last injection). Patients enrolled into the study not progressing at the time of study stop, and who agree to stay on LAN therapy (i.e. OL Treatment Period) receive the study active treatment until evidence of disease progression (based on local radiological assessment then confirmed centrally), development of unacceptable toxicity, or premature withdrawal for any reason or up a maximum of 18 months after the last patient randomized. After disease progression patients are followed for survival, QoL and all subsequent anticancer treatments in the OL Follow-up period up to the end of the study (i.e up to 18 months after the last patient randomized).

ELIGIBILITY:
Inclusion Criteria:

* Have metastatic and/or unresectable pathologically confirmed well-differentiated, typical or atypical neuroendocrine tumor of the bronchopulmonary
* Histologic evidence of Well differentiated Neuroendocrine tumors (NETs) of the bronchopulmonary (typical and atypical according to the World Health Organisation (WHO criteria), evaluated locally)
* Has a mitotic index <2 mitoses/2 mm2 for typical carcinoid (TC) and <10 mitoses/2 mm2 and/or foci of necrosis for atypical carcinoid (AC)
* At least one measurable lesion of the disease on imaging (CT or MRI; RECIST 1.1)
* Positive Somatostatin receptors (SSTR) imaging

Exclusion Criteria:

* Poorly differentiated or high grade carcinoma, or patients with neuroendocrine tumors not of bronchopulmonary origin
* Has been treated with a Somatostatin analog (SSA) at any time prior to randomization, except if that treatment was for less than 15 days (e.g. peri-operatively) of short acting SSA or one dose of long acting SSA and the treatment was received more than 6 weeks prior to randomization
* Has been treated with Peptide receptor radionuclide therapy (PRRT) at any time prior to randomization
* Has been treated with more than two lines of cytotoxic chemotherapy or molecular targeted therapy or interferon for bronchopulmonary NET

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (57):
- United States (14):
  - Arizona Oncology Associates, Tucson, Arizona
  - VA Greater Los Angeles, Los Angeles, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Ochsner Medical Center, New Orleans, Louisiana
  - Dana-Farber Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Science Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Oncology, Dallas, Texas
  - Texas Oncology-Forth Worth, Fort Worth, Texas
- Austria (2):
  - AKH und Med. University Vienna Allg Krankenhaus Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Canada (6):
  - Tom Baker Cancer Center, Calgary, Alberta
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon
  - Cancer Care of Manitoba, Winnipeg
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - NET-Centre, Rigshospitalet, Copenhagen
- France (7):
  - Centre Oscar Lambret, Lille
  - Hôpital Edouard Herriot, Lyon
  - CLLC, Institut Paoli Calmettes, Marseille
  - Institut du Cancer de Montpellier (ICM) Val d'Aurelle, Montpellier
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Centre René Gauducheau ICO institut de Cancerologie de l'Ouest, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitätsklinikum Essen (AöR), Essen
  - Johann Wolfgang Goethe-Universitätsklinikum Frankfurt, Frankfurt
- Italy (5):
  - Universita di Genova, Genova
  - Insituti Scientifico Romagnolo per lo Studio e la cura dei Tumori (IRST), Meldola
  - Azienda Ospedaliera Antonio Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria di Perugia Santa Maria della Misericordia, Perugia
  - Insittuto Clinico Humanitas, Rozzano
- Netherlands (2):
  - Antoni van Leeuwenhoek, Amsterdam
  - Maastricht University Medical Center, Maastricht
- Poland (5):
  - Zakladu Medycyny Nuklearne i Endokrynologii Onkologicznej, Gliwice
  - University Center of Ophtalmology & Oncology, Katowice
  - Szpital Uniwersytecki W, Krakow
  - Szpital Kliniczny im. H. Święcickiego U.M., Poznan
  - GAMMED, Warsaw
- Spain (4):
  - Hospital Universitari, Vall d'Hebron, Barcelona
  - University Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (6):
  - Cancer Center, Beatson Oncology, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Royal Free Hospital, London
  - King's College Hospital, London
  - Christie Hospital, Manchester
  - Churchill Hospital, Oxford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 37 investigation sites in 10 countries in North America and Europe between 06 March 2017 and 28 February 2020 in adult subjects with well differentiated, metastatic and/or unresectable, typical or atypical bronchopulmonary (BP) neuroendocrine tumours (NETs) who did not require somatostatin analogue (SSA) treatment for symptom control.
Pre-assignment Details: This study consisted of two phases: the double-blind phase, and the open-label phase. 77 subjects were randomised to receive study treatment until disease progression, unacceptable toxicity, withdrawal for any reason, or up to 18 months after the last subject was randomised. Subjects were randomised 2:1 to either lanreotide autogel/depot 120 milligrams (mg) plus best supportive care (BSC) every 28 days (Q4 weeks) or placebo plus BSC Q4 weeks.
Groups:
- Lanreotide: Subjects received deep subcutaneous (SC) injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. Following protocol amendment #5 (28 Jan 2019), all ongoing subjects in the double-blind phase, who had not yet progressed (assessed locally and confirmed centrally) were offered to enter the open-label treatment phase and continue to receive deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. If a subject progressed during the double-blind phase or open-label treatment phase they entered the open-label follow-up phase. The follow-up phase ended at the same time as the open-label treatment phase (18 months after the last subject randomised).
- Placebo: Subjects received deep SC injections of placebo (saline solution 0.9%) Q4 weeks plus BSC in the double-blind phase. Following protocol amendment #5 (28 Jan 2019), all ongoing subjects in the double-blind phase, who had not yet progressed (assessed locally and confirmed centrally) were offered to enter the open-label treatment phase and receive deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. If a subject progressed during the open-label treatment phase they entered the open-label follow-up phase. The follow-up phase ended at the same time as the open-label treatment phase (18 months after the last subject randomised).
Period: Double-blind Phase
Arm/Group | Lanreotide | Placebo
Started | 51 | 26
Completed (Completers are subjects who complete the double-blind phase of the study or die.) | 41 | 21
Not Completed | 10 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Disease Progression | 5 | 2
Period: Open-label Treatment Phase
Arm/Group | Lanreotide | Placebo
Started (Prior to protocol amendment #5, subjects qualified for the option to continue into the open-label treatment phase if they met the following additional inclusion criteria: * Subjects have central review confirmed/documented disease progression; * There was a request from the subject to receive open-label lanreotide plus BSC; * Subjects were randomized in the placebo plus BSC arm. Following protocol amendment #5, the open-label treatment phase remained optional for all subjects.) | 21 | 19
Completed (Completers are subjects who complete the open-label treatment phase of the study or die.) | 1 | 6
Not Completed | 20 | 13
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Disease Progression | 1 | 2
Not completed — Study Termination by the Sponsor | 18 | 9
Not completed — Other | 1 | 0
Period: Open-label Follow-up Phase
Arm/Group | Lanreotide | Placebo
Started (Inclusive of subjects who progressed during the double-blind phase or open-label treatment phase.) | 18 | 8
Completed | 0 | 0
Not Completed | 18 | 8
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study Termination by the Sponsor | 6 | 4
Not completed — Other | 8 | 1

BASELINE CHARACTERISTICS:
Population: The intention to treat (ITT) population included all randomised subjects. Subjects were analysed as randomised, regardless of the treatment received.
Groups:
- Lanreotide: Subjects received deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. Following protocol amendment #5 (28 Jan 2019), all ongoing subjects in the double-blind phase, who had not yet progressed (assessed locally and confirmed centrally) were offered to enter the open-label treatment phase and receive deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. If a subject progressed during the double-blind phase or open-label treatment phase they entered the open-label follow-up phase. The follow-up phase ended at the same time as the open-label treatment phase (18 months after the last subject randomised).
- Total: Total of all reporting groups
Arm/Group | Lanreotide | Placebo | Total
Number analyzed (Participants) | 51 | 26 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (11.94) | 65.8 (13.89) | 66.2 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 28 | 14 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 0
  Ethnicity: Not Hispanic or Latino | 9 | 4 | 13
  Ethnicity: Missing | 42 | 22 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 3 | 0 | 3
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 1 | 0 | 1
  Race: White | 35 | 19 | 54
  Race: More than one race | 0 | 0 | 0
  Race: Missing | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-Free Survival (PFS) Time in Subjects Randomised to Lanreotide in the Double-Blind Phase or Open-Label Treatment Phase, Assessed by Central Review
Description: PFS for subjects randomised in the lanreotide group, assessed by central review using Response Evaluation Criteria In Solid Tumours Version 1.1 (RECIST v1.1) criteria every 12 weeks, defined as the time from randomisation to disease progression or death from any causes during either the double-blind phase, or the open-label treatment phase. The distribution of PFS times were estimated using the Kaplan-Meier product limit method.
Time Frame: Up to a maximum of 33 months
Population: The ITT population included all randomised subjects. Subjects were analysed as randomised, regardless of the treatment received. One subject randomised to lanreotide should have been censored in the PFS analysis treatment for discontinuation for toxicity or other reasons, however the baseline central radiological assessment was performed prior to the randomisation date, therefore the subject was excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Overall Study: Lanreotide: Subjects received deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. Following protocol amendment #5 (28 Jan 2019), all ongoing subjects in the double-blind phase, who had not yet progressed (assessed locally and confirmed centrally) were offered to enter the open-label treatment phase and continue to receive deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. If a subject progressed during the double-blind phase or open-label treatment phase they entered the open-label follow-up phase. The follow-up phase ended at the same time as the open-label treatment phase (18 months after the last subject randomised).
Arm/Group | Overall Study: Lanreotide
Number analyzed (Participants) | 50
months | 16.6 [11.3 to 21.9]

2. Secondary Outcome: Median PFS Time in the Double-Blind Phase, Assessed by Central Review
Description: PFS was assessed by central review using RECIST v1.1 criteria every 12 weeks, defined as the time from randomisation to disease progression or death from any causes during the double-blind phase. The distribution of PFS times were estimated using the Kaplan-Meier product limit method.
Time Frame: Up to a maximum of 15 months
Population: The ITT population included all randomised subjects. Subjects were analysed as randomised, regardless of the treatment received. One subject in the double-blind phase: lanreotide arm should have been censored in the PFS analysis for treatment discontinuation for toxicity or other reasons, however the baseline central radiological assessment was performed prior to the randomisation date, therefore the subject was excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Double-Blind Phase: Lanreotide: Subjects received deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. Following protocol amendment #5 (28 Jan 2019), all ongoing subjects in the double-blind phase, who had not yet progressed (assessed locally and confirmed centrally) were offered to enter the open-label treatment phase and continue to receive deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. If a subject progressed during the double-blind phase they entered the open-label follow-up phase.
- Double-Blind Phase: Placebo: Subjects received deep SC injections of placebo (saline solution 0.9%) Q4 weeks plus BSC in the double-blind phase. Following protocol amendment #5 (28 Jan 2019), all ongoing subjects in the double-blind phase, who had not yet progressed (assessed locally and confirmed centrally) were offered to enter the open-label treatment phase and receive deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC.
Arm/Group | Double-Blind Phase: Lanreotide | Double-Blind Phase: Placebo
Number analyzed (Participants) | 50 | 26
months | 16.6 [11.3 to 21.9] | 13.6 [8.3 to NA] — Upper confidence interval not calculable due to insufficient progression events.
Statistical Analysis 1: Comparison: Double-Blind Phase: Lanreotide vs Double-Blind Phase: Placebo; The hazard ratio and the 95% confidence interval (CI) were estimated using a Cox proportional hazards model, stratified for interactive web response system (IWRS) tumour subtype (typical versus [vs] atypical) using the exact method for ties. P-value of stratified log rank test comparing lanreotide to placebo with strata based on the IWRS tumour subtype (typical vs atypical) stratification factor; Test type: Superiority; p = 0.866, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.48 to 1.95]

3. Secondary Outcome: Median PFS Time in the Double-Blind Phase, Assessed by Local Review
Description: PFS was assessed by local review using RECIST v1.1 criteria every 12 weeks, defined as the time from randomisation to disease progression or death from any causes during the double-blind phase. The distribution of PFS times were estimated using the Kaplan-Meier product limit method.
Time Frame: Up to a maximum of 15 months
Population: The ITT population included all randomised subjects. Subjects were analysed as randomised, regardless of the treatment received. Two subjects should have been censored in the PFS analysis, however the baseline central radiological assessment was performed prior to the randomisation date, therefore the subjects were excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Double-Blind Phase: Lanreotide | Double-Blind Phase: Placebo
Number analyzed (Participants) | 50 | 25
months | 14.1 [11.1 to NA] — Upper confidence interval not calculable due to insufficient progression events. | 13.6 [8.3 to NA] — Upper confidence interval not calculable due to insufficient progression events.
Statistical Analysis 1: Comparison: Double-Blind Phase: Lanreotide vs Double-Blind Phase: Placebo; The hazard ratio and the 95% CI were estimated using a Cox proportional hazards model, stratified for IWRS tumour subtype (typical vs atypical) using the exact method for ties. P-value of stratified log rank test comparing lanreotide to placebo with strata based on the IWRS tumour subtype (typical vs atypical) stratification factor; Test type: Superiority; p = 0.837, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.48 to 1.88]

4. Secondary Outcome: Objective Response Rate (ORR) in the Double-Blind Phase
Description: ORR was assessed by central review and local review using RECIST v1.1 criteria every 12 weeks, defined as the percentage of subjects who achieved a best overall response of complete response or partial response in the double-blind phase.
Time Frame: Up to a maximum of 15 months
Population: The ITT population included all randomised subjects. Subjects were analysed as randomised, regardless of the treatment received. Two subjects were excluded from the analysis as they had no best response recorded in the raw data.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Double-Blind Phase: Lanreotide | Double-Blind Phase: Placebo
Number analyzed (Participants) | 50 | 25
Percentage of subjects
  Central review | 14.00 [5.82 to 26.74] | 0.00 [0.00 to 13.72]
  Local review | 6.00 [1.25 to 16.55] | 4.00 [0.10 to 20.35]
Statistical Analysis 1: Comparison: Double-Blind Phase: Lanreotide vs Double-Blind Phase: Placebo; The treatment difference compares lanreotide to placebo (central review). The 95% exact unconditional CI was used for ORR difference; Test type: Other; Percentage difference = 14.00, 95% CI 2-sided [-10.97 to 37.86]
Statistical Analysis 2: Comparison: Double-Blind Phase: Lanreotide vs Double-Blind Phase: Placebo; The treatment difference compares lanreotide to placebo (local review). The 95% exact unconditional CI was used for ORR difference; Test type: Other; Percentage difference = 2.00, 95% CI 2-sided [-22.69 to 26.53]

5. Secondary Outcome: Time to Treatment Failure (TTF) in the Double-Blind Phase
Description: TTF was defined as the time from randomisation to disease progression using RECIST v1.1, death, consent withdrawn, an adverse event, protocol deviations, lost to follow-up, the appearance of carcinoid syndrome or other hormone related syndrome necessitating the initiation of SSAs (rescue octreotide and/or long-acting release SSA), or initiation of anticancer treatment in the double-blind phase. The distribution of TTF times were estimated using the Kaplan-Meier product limit method.
Time Frame: Up to a maximum of 15 months
Population: The ITT population included all randomised subjects. Subjects were analysed as randomised, regardless of the treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Double-Blind Phase: Lanreotide | Double-Blind Phase: Placebo
Number analyzed (Participants) | 51 | 26
months | 13.3 [5.6 to 14.1] | 9.8 [5.4 to 13.6]
Statistical Analysis 1: Comparison: Double-Blind Phase: Lanreotide vs Double-Blind Phase: Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.582, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.50 to 1.50]

6. Secondary Outcome: Mean Change From Baseline in the Biomarker Chromogranin A (CgA) in the Double-Blind Phase and Open-Label Treatment Phase
Description: Blood samples were collected to determine plasma CgA. Baseline was defined as the last non-missing measurement collected prior to the first dose of study treatment (lanreotide). The x of upper limit of normal (ULN) was calculated as raw value/ULN.
Time Frame: Baseline, Weeks 8, 12, 24, and 48, and post-treatment in the double-blind phase (a maximum of 15 months); Baseline, Weeks 12, 24, and 48, and post-treatment in the the open-label treatment phase (a maximum of 33 months)
Population: Double-blind phase: The ITT population included all randomised subjects with non-missing measurements. Subjects were analysed as randomised, regardless of the treatment received. Open-label phase: The open-label ITT population included all ITT subjects with non-missing measurements entering the open-label phase who received at least one injection of lanreotide autogel/depot in the open-label phase.
Measure: Mean (Standard Deviation); unit: x of ULN
Groups:
- Open-Label Treatment Phase: All Subjects: Subjects received deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. Following protocol amendment #5 (28 Jan 2019), all ongoing subjects in the double-blind phase, who had not yet progressed (assessed locally and confirmed centrally) were offered to enter the open-label treatment phase and receive deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. If a subject progressed during the open-label treatment phase they entered the open-label follow-up phase.
Arm/Group | Double-Blind Phase: Lanreotide | Double-Blind Phase: Placebo | Open-Label Treatment Phase: All Subjects
Number analyzed (Participants) | 38 | 22 | 33
x of ULN
  Week 8: number analyzed (Participants) | 38 | 22 | 0
  Week 8 | -213.63 (1293.111) | 0.09 (2.578) |
  Week 12: number analyzed (Participants) | 38 | 20 | 33
  Week 12 | -214.49 (1344.401) | 5.73 (15.519) | -28.27 (149.110)
  Week 24: number analyzed (Participants) | 33 | 19 | 30
  Week 24 | -3.42 (14.122) | 60.41 (193.327) | -1.42 (8.338)
  Week 48: number analyzed (Participants) | 24 | 11 | 7
  Week 48 | -4.07 (8.066) | 1.24 (2.969) | -1.66 (0.925)
  Post-treatment: number analyzed (Participants) | 33 | 14 | 31
  Post-treatment | 12.22 (64.053) | 160.11 (596.759) | -31.59 (167.515)

7. Secondary Outcome: Percentage of Subjects With a Decrease of CgA ≥30% From Baseline at Week 8 in the Double-Blind Phase and Open-Label Treatment Phase
Description: Measured in subjects with an elevated CgA at baseline (≥2 x ULN). Blood samples were collected to determine plasma CgA. Baseline was defined as the last non-missing measurement collected prior to the first dose of study treatment (lanreotide).
Time Frame: Baseline and Week 8 in the double-blind phase; Baseline and Week 8 in the open-label treatment phase
Population: Double-blind phase: The ITT population included all randomised subjects with non-missing measurements and elevated CgA at Baseline. Subjects were analysed as randomised, regardless of the treatment received. Open-label phase: The open-label ITT population included all ITT subjects with non-missing measurements and elevated CgA at Baseline entering the open-label phase who received at least one injection of lanreotide autogel/depot in the open-label phase.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Double-Blind Phase: Lanreotide | Double-Blind Phase: Placebo | Open-Label Treatment Phase: All Subjects
Number analyzed (Participants) | 30 | 13 | 19
percentage of subjects | 63.3 [43.9 to 80.1] | 7.7 [0.2 to 36.0] | 73.7 [48.8 to 90.9]

8. Secondary Outcome: Mean Changes From Baseline in Quality of Life (QoL), as Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) Global Health Status/QoL Score
Description: The EORTC QLQ-C30 (V3.0) consisted of 30 questions. The final 2 questions were related to global health status/QoL, with responses requested on a 7-point scale from 1 ('Very poor') to 7 ('Excellent'). The global health status/QoL scale ranges in score from 0 to 100. A high score for the global health status/QoL scale represents a high QoL, thus, an increase in score represents an increase in QoL. 95% Clopper-Pearson confidence intervals were estimated using the exact method for binomial distributions. Baseline was defined as the last non-missing measurement collected prior to the first dose of study treatment (lanreotide).
Time Frame: Baseline and post-treatment in the double-blind phase (a maximum of 15 months); Baseline and post-treatment in the open-label treatment phase (a maximum of 33 months)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Double-Blind Phase: Lanreotide | Double-Blind Phase: Placebo | Open-Label Treatment Phase: All Subjects
Number analyzed (Participants) | 25 | 3 | 34
score on a scale | -2.7 (18.27) | -19.4 (17.33) | 0.0 (19.67)

9. Secondary Outcome: Percentage of Subjects Who Experienced QoL Deterioration
Description: QoL deterioration was defined by a decrease from baseline in EORTC QLQ-C30 Global Health Status/QoL Score of at least 10 points. The EORTC QLQ-C30 (V3.0) consisted of 30 questions. The final 2 questions were related to global health status/QoL, with responses requested on a 7-point scale from 1 ('Very poor') to 7 ('Excellent'). The global health status/QoL scale ranges in score from 0 to 100. A high score for the global health status/QoL scale represents a high QoL, thus, an increase in score represents an increase in QoL. 95% Clopper-Pearson confidence intervals were estimated using the exact method for binomial distributions. Baseline was defined as the last non-missing measurement collected prior to the first dose of study treatment (lanreotide).
Time Frame: as for outcome 8
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Double-Blind Phase: Lanreotide | Double-Blind Phase: Placebo | Open-Label Treatment Phase: All Subjects
Number analyzed (Participants) | 25 | 3 | 34
percentage of subjects | 32.0 [14.9 to 53.5] | 66.7 [9.4 to 99.2] | 23.5 [10.7 to 41.2]

10. Secondary Outcome: Mean Changes From Baseline in Urinary 5-hydroxyindoleacetic Acid (5-HIAA) Levels in the Double-Blind Phase and Open-Label Treatment Phase
Description: Measured in subjects with an elevated 5-HIAA at baseline (≥2 x ULN). The assessment of urinary 5-HIAA required subjects to collect their urine for the 24 hour period prior to the study visit. Baseline was defined as the last non-missing measurement collected prior to the first dose of study treatment (lanreotide). The x of ULN was calculated as raw value/ULN.
Time Frame: as for outcome 6
Population: Double-blind phase: The ITT population included all randomised subjects with non-missing measurements and elevated 5-HIAA at baseline. Subjects were analysed as randomised, regardless of the treatment received. Open-label phase: The open-label ITT population included all ITT subjects with non-missing measurements and elevated 5-HIAA at baseline entering the open-label phase who received at least one injection of lanreotide autogel/depot in the open-label phase.
Measure: Mean (Standard Deviation); unit: x of ULN
Arm/Group | Double-Blind Phase: Lanreotide | Double-Blind Phase: Placebo | Open-Label Treatment Phase: All Subjects
Number analyzed (Participants) | 7 | 4 | 3
x of ULN
  Week 8: number analyzed (Participants) | 7 | 4 | 0
  Week 8 | -2.90 (5.368) | 2.78 (4.215) |
  Week 12: number analyzed (Participants) | 5 | 3 | 2
  Week 12 | 0.21 (1.904) | 5.38 (4.342) | -0.47 (1.886)
  Week 24: number analyzed (Participants) | 5 | 2 | 3
  Week 24 | 0.15 (3.041) | -1.40 (2.734) | -4.84 (10.019)
  Week 48: number analyzed (Participants) | 4 | 1 | 1
  Week 48 | -3.00 (8.900) | 1.13 (NA) — Standard deviation was not calculable as only 1 subject was analysed. | -2.47 (NA) — Standard deviation was not calculable as only 1 subject was analysed.
  Post-treatment: number analyzed (Participants) | 5 | 2 | 2
  Post-treatment | -1.27 (7.007) | -5.13 (11.597) | 0.60 (3.583)

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last study treatment administration/early termination, approximately 33 months
Description: The safety population included all subjects who received at least one injection of study treatment. Subjects were analysed as treated.
Groups:
- Open-Label Treatment Phase: Subjects received deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. Following protocol amendment #5 (28 Jan 2019), all ongoing subjects in the double-blind phase, who had not yet progressed (assessed locally and confirmed centrally) were offered to enter the open-label treatment phase and receive deep SC injections of lanreotide autogel/depot 120 mg Q4 weeks plus BSC. If a subject progressed during the open-label treatment phase they entered the open-label follow-up phase.
- Open-Label Follow-Up Phase: If the subject received lanreotide autogel/depot and progressed during the double-blind phase or open-label treatment phase, the subject entered the follow-up phase of the open-label treatment phase and was followed for QoL/survival and all subsequent anticancer treatments received. No intervention was received in the open-label follow-up phase.
Arm/Group | Double-Blind Phase: Lanreotide | Double-Blind Phase: Placebo | Open-Label Treatment Phase | Open-Label Follow-Up Phase
All-Cause Mortality (participants affected / at risk) | 2/51 | 0/26 | 0/40 | 7/26
Serious Adverse Events (participants affected / at risk) | 10/51 | 7/26 | 1/40 | 0/26
Other Adverse Events (participants affected / at risk) | 48/51 | 25/26 | 26/40 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Phase: Lanreotide (N=51) | Double-Blind Phase: Placebo (N=26) | Open-Label Treatment Phase (N=40) | Open-Label Follow-Up Phase (N=26)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Phase: Lanreotide (N=51) | Double-Blind Phase: Placebo (N=26) | Open-Label Treatment Phase (N=40) | Open-Label Follow-Up Phase (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (3) | 2 (3) | 3 (4) | 0 (0)
Carcinoid syndrome (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 5 (14) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (21) | 5 (8) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 2 (4) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (9) | 4 (4) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 32 (61) | 8 (12) | 9 (13) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 7 (12) | 2 (2) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycogenic acanthosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (17) | 4 (4) | 3 (5) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Steatorrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (8) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 11 (19) | 5 (11) | 2 (10) | 0 (0)
Chest pain (General disorders) | 2 (5) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 13 (20) | 10 (10) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 4 (5) | 1 (1) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 5 (10) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Xerosis (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (6) | 4 (4) | 2 (4) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 3 (6) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood albumin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Intestinal transit time increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 4 (5) | 3 (3) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7) | 6 (7) | 3 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 4 (11) | 1 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2) | 2 (2) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 8 (15) | 2 (2) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 4 (4) | 4 (5) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract discomfort (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3) | 2 (4) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 4 (4) | 2 (3) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2) | 1 (2) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Melanoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 5 (14) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contrast media reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 3 (3) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mediastinal fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The majority of subjects who entered the open-label treatment phase were withdrawn due to study termination by the sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT02683941/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT02683941/SAP_001.pdf